CLINICAL TRIAL: NCT04805216
Title: A Single-centre, Observational Study to Evaluate Immune Response to Covid-19 Vaccines in Immunocompromised Patients With Haematological Disorders
Brief Title: Covid-19 Vaccine Response in Immunocompromised Haematology Patients
Acronym: COVAC-IC
Status: Completed | Type: Observational
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Collaborators: University Hospitals of North Midlands NHS Trust Charity (Unknown); Staffordshire University (Other)
Responsible Party: Sponsor
Other Study IDs: 3025
Record Dates: First submitted 2021-03-12; First posted 2021-03-18 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2022-02

CONDITIONS: Covid19; Haematological Disorders; Immune Suppression
MeSH Terms: conditions — COVID-19; Hematologic Diseases | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immunocompromised patients (study group): People who are likely to have a suppressed immunity due to their haematological disorder or its treatment
  Interventions: Procedure: Blood test
- Immunocompetent volunteers (control group): People without suppressed immunity
  Interventions: Procedure: Blood test

INTERVENTIONS:
Procedure: Blood test — Participants will have blood tests at baseline (nearest 30 day incremental time point after 2nd dose of Covid-19 vaccine, +/- 7 days):
  * T, B & NK cells
  * Full Blood Count and differential
  * Serum Immunoglobulins
  * Antibodies against VZV, CMV, Rubella
  * Quantiferon assay (T-Cell response)
  * Covid antibody assay (LIAISON® SARS-CoV-2 S1/S2 IgG quantitative assay)
  Participants will have blood tests during follow up (after second dose of Covid-19 vaccine) with a window of +/- 7 days:
  * Blood test 2 - performed at the next 30 day time point (Covid antibody assay)
  * Blood test 3 - performed at the next 30 day time point (Covid antibody assay and quantiferon* if final blood test)
  * Blood test 4 (optional) - performed at the next 30 day time point (Covid antibody assay)
  * Blood test 5 (optional) - performed at the next 30 day time point (Covid antibody assay and quantiferon* if final blood test)
    * Quantiferon assay will be only be performed where possible.

SUMMARY:
The UK Medicine and Healthcare products Regulatory Agency (MHRA) granted temporary authorisation to three Covid-19 vaccines in December 2020 and January 2021.

These vaccinations include:

* Covid-19 mRNA BNT162b2 vaccine (Pfizer-BioNtech vaccine);
* ChAdOx1-S vaccine (Astra Zeneca vaccine);
* Covid-19 mRNA vaccine (Moderna vaccine).

Any other Covid-19 vaccines approved for use by the MHRA in immunocompromised and immunocompetent patients are to be included in this study. The above vaccines have received temporary authorisation after placebo-controlled phase 3 studies confirmed their safety and efficacy in over 100,000 volunteers. People who were immunocompromised or were receiving chemotherapy, radiotherapy or immunoglobulin treatment were excluded from these studies. Safety, efficacy, and durability of antibody response in these studies has been assessed for up to 14 weeks only. These vaccines are being rolled out in the UK and have been recommended for use for immunosuppressed individuals including patients undergoing chemotherapy, immunotherapy, radiotherapy, and those who have undergone stem cell transplantation. Though the MHRA has approved vaccination for immunocompromised patients there is no published evidence to confirm safety and efficacy in these patients. The durability of antibody response and whether this is affected by concurrent chemotherapy, immunotherapy, radiotherapy treatment is also unknown.

This observational study aims to evaluate the immune response to Covid-19 vaccines in haematology patients who have immune suppression either due to disease, treatment, or both. The investigators plan to measure Anti-SARS-COV2 IgG antibody levels at 3-5 time points 30 days apart after patients have received their 2nd dose of Covid-19 vaccine. The investigators will also collect any adverse events reported by patient including Covid-19 infection or disease after vaccination.

The study plans to recruit 50 haematology patients who are clinically assessed by a haematologist as immunosuppressed due to their disease, treatment, or both. The study also plans to recruit 30 healthy (immunocompetent) volunteers who would be the control group for comparison of antibody response and durability.

ELIGIBILITY:
Inclusion Criteria (Immunocompromised Haematology Patients)

* Aged 18 years and over;
* Has one or more haematological disorder(s) with compromised immunity or currently receiving or recently treated (within previous 3 months of the screening appointment date) with immunosuppressive therapy, chemotherapy, radiotherapy or stem cell transplantation;
* Has had at least 2 doses of Covid-19 vaccine;
* Willing and able to give fully informed consent;
* Willing and able to comply with the study procedures;
* Anticipated life expectancy of over 6 months.

Exclusion Criteria (Immunocompromised Haematology Patients)

* Has declined or does not wish to have Covid-19 vaccine;
* Is receiving regular IV Immunoglobulins for immunodeficiency;
* Is taking part in an interventional Covid-19 vaccine study;
* Ineligible* for Covid-19 vaccine;
* Non-English speaker where translation facilities are insufficient to guarantee informed consent.

  * Ineligible for health reasons and/or as per Government prioritisation of vaccinations

Inclusion Criteria (Control group - Immunocompetent Volunteers)

* Aged 18 years and over;
* Is immunocompetent;
* Has had at least 2 doses of Covid-19 vaccine;
* Anticipated life expectancy of over 6 months;
* Willing and able to give fully informed consent;
* Willing and able to comply with the study procedures.

Exclusion Criteria (Control group - Immunocompetent Volunteers)

* Has declined or does not wish to have Covid-19 vaccine;
* Has comorbidity known to result in immune suppression;
* Has received treatment (within previous 12 months of the screening appointment) with immunosuppressive therapy, chemotherapy, radiotherapy or stem cell transplantation;
* Is taking part in an interventional Covid-19 vaccine study;
* Ineligible for Covid-19 vaccine*;
* Non-English speaker where translation facilities are insufficient to guarantee informed consent.

  * Ineligible for health reasons and/or as per Government prioritisation of vaccinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 Immunocompromised haematology patients (also referred to as the "study group") and 30 Immunocompetent, healthy volunteers (also referred to as the "control group")
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Anti-SARS-COV2 IgG antibodies in immunocompromised haematology patients compared to immunocompetent controls over a 4 month period | Nearest 30 day time point after 2nd dose Covid-19 vaccination (baseline) and every 30 days (3-5 follow-up time points) after 2nd dose of Covid-19 vaccination (+/- 7 days)
  Anti-SARS-COV2 IgG antibodies
Duration of Anti-SARS-COV2 IgG antibody response in immunocompromised haematology patients compared to immunocompetent controls over a 4 month period | Nearest 30 day time point after 2nd dose Covid-19 vaccination (baseline)
  Duration of Anti-SARS-COV2 IgG antibody response
Duration of Anti-SARS-COV2 IgG antibody response in immunocompromised haematology patients compared to immunocompetent controls over a 4 month period | 30 days follow-up (+/- 7 days)
  Duration of Anti-SARS-COV2 IgG antibody response
Duration of Anti-SARS-COV2 IgG antibody response in immunocompromised haematology patients compared to immunocompetent controls over a 4 month period | 60 days follow-up (+/- 7 days)
  Duration of Anti-SARS-COV2 IgG antibody response
Duration of Anti-SARS-COV2 IgG antibody response in immunocompromised haematology patients compared to immunocompetent controls over a 4 month period | 90 days follow-up (+/- 7 days) - optional
  Duration of Anti-SARS-COV2 IgG antibody response
Duration of Anti-SARS-COV2 IgG antibody response in immunocompromised haematology patients compared to immunocompetent controls over a 4 month period | 120 days follow-up (+/- 7 days) - optional
  Duration of Anti-SARS-COV2 IgG antibody response

SECONDARY OUTCOMES:
Correlation in antibody response with patient gender | From recruitment until up to 120 days follow-up (+/- 7 days)
  Gender and anti-SARS-Cov-2 IgG antibodies
Correlation in antibody response with patient ethnicity | From recruitment until up to 120 days follow-up (+/- 7 days)
  Ethnicity and anti-SARS-Cov-2 IgG antibodies
Correlation in antibody response with patient haematological disorder | From recruitment until up to 120 days follow-up (+/- 7 days)
  Haematological disorder and anti-SARS-Cov-2 IgG antibodies
Correlation in antibody response with patient age | From recruitment until up to 120 days follow-up (+/- 7 days)
  Age and anti-SARS-Cov-2 IgG antibodies
Correlation in antibody response with patient treatment | From recruitment until up to 120 days follow-up (+/- 7 days)
  Treatment and anti-SARS-Cov-2 IgG antibodies
Correlation in antibody response with patient Covid-19 vaccine type | From recruitment until up to 120 days follow-up (+/- 7 days)
  Covid-19 vaccine type and anti-SARS-Cov-2 IgG antibodies
Correlation in antibody response with patient pre-vaccine immunological parameters | From recruitment until up to 120 days follow-up (+/- 7 days)
  Pre-vaccine immunological parameters and anti-SARS-Cov-2 IgG antibodies
Adverse events associated with the first and second dose of a Covid-19 vaccination, reported by the study group and control group | From recruitment until up to 120 days follow-up (+/- 7 days)
  Any participant-reported adverse events via baseline CRF
PCR positive Covid-19 infections reported by the study group and control group | From recruitment until up to 120 days follow-up (+/- 7 days, as reported during this time frame)
  Patient reported Covid-19 PCR test via CRF, if performed on participant (routine PCR testing is not part of study)
T-Cell response after second dose Covid-19 vaccination in immunocompromised haematology patients compared to immunocompetent controls over a 4 month period | From recruitment and at 60 or 90 days follow-up (+/- 7 days)
  T-Cell cytokine response to 2nd dose Covid-19 vaccine
Duration of T-Cell response after second dose Covid-19 vaccination in immunocompromised haematology patients compared to immunocompetent controls over a 4 month period | From recruitment and at 60 or 90 days follow-up (+/- 7 days)
  Duration of T-Cell cytokine response to 2nd dose Covid-19 vaccine

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, United Kingdom

IPD SHARING:
Plan to Share IPD: No